CLINICAL TRIAL: NCT07321015
Title: An Exploratory Single-Arm Study of Maintenance Fluzoparib in Platinum-Sensitive, Advanced Triple-Negative Breast Cancer Patients With BRCA1/2 Mutation or Wild-Type BRCA
Brief Title: A Single-Arm Phase Ⅱ Study of Fluzoparib Maintenance in Platinum-sensitive Advanced Triple-Negative Breast Cance
Acronym: Fzp-MA-TNBC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK20250453
Record Dates: First submitted 2025-12-02; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Platinum-sensitive; TNBC, Triple Negative Breast Cancer; BRCA1/2 Mutation or Not
Keywords: TNBC; Platinum-sensitive; Maintenance Therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib Maintenance Until Disease Progression or Intolerable Toxicity (Experimental): Patients with advanced triple-negative breast cancer who have achieved at least stable disease (SD) or partial response (PR) after ≥2 prior lines of therapy including a platinum-based regimen will receive fluzoparib 150 mg orally twice daily on days 1-28 of each 28-day cycle. Treatment continues until disease progression, unacceptable toxicity, withdrawal of consent, or death. Dose interruptions or reductions (to 100 mg BID or 50 mg BID) are allowed for predefined toxicities. No concurrent anticancer therapy is permitted. Efficacy assessments (CT/MRI) will be performed every 6 weeks (2 cycles) from the first dose. Exploratory biomarkers (PD-L1, TILs, CD4/8, cytokines) will be collected optionally for subgroup analyses.
  Interventions: Drug: Fluzoparib Monotherapy

INTERVENTIONS:
Drug: Fluzoparib Monotherapy — Fluzoparib is an oral poly (ADP-ribose) polymerase (PARP) inhibitor supplied as 50 mg capsules. Participants take 150 mg twice daily (total 300 mg/day) on days 1-28 of each 28-day cycle. Doses should be swallowed whole with water, approximately 12 hours apart, at approximately the same times each day. Treatment continues until disease progression, unacceptable toxicity, withdrawal of consent, or death. Dose interruptions or reductions (stepwise to 100 mg BID or 50 mg BID) are allowed for haematological or non-haematological toxicities graded ≥3 or as clinically indicated. No concurrent anticancer therapy is permitted during fluzoparib maintenance.

SUMMARY:
Breast cancer is the most common malignancy in women; approximately 5-10% are hereditary, with 14% of triple-negative breast cancers (TNBC) harboring BRCA mutations. BRCA1/2 are essential for homologous recombination repair of DNA double-strand breaks, whereas PARP mediates base-excision repair of single-strand breaks. PARP inhibitors (PARPi) exploit synthetic lethality to selectively eliminate BRCA-deficient tumor cells. Olaparib and talazoparib have demonstrated superior PFS and ORR versus chemotherapy in BRCA-mutated, HER2-negative advanced breast cancer, leading to FDA approval. In ovarian cancer, PARPi maintenance improves overall survival, with consistent benefits observed in Asian populations. The domestically developed PARPi fluzoparib, engineered with a trifluoromethyl moiety for enhanced stability and tissue penetration, showed in the phase III FABULOUS trial a median PFS of 6.7 vs 3.0 months and an ORR of 43.6% vs 23.3% compared with chemotherapy in gBRCA-mutated, HER2-negative breast cancer, with manageable safety. Data remain limited in Chinese patients and those with BRCA wild-type disease. This study aims to evaluate the efficacy and safety of fluzoparib maintenance monotherapy in advanced TNBC patients-either BRCA1/2-mutated or wild-type-who have derived clinical benefit from prior platinum-based therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years (inclusive) at the time of informed consent.
2. Histologically confirmed triple-negative breast cancer (TNBC; ER <1%, PR <1%, HER2-negative).
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Received ≥2 prior lines of systemic therapy, including a platinum-based regimen (single-agent or combination); must have achieved partial response (PR) or stable disease (SD) during or after that platinum-based treatment.
5. Platinum-sensitive disease defined as: Objective response (complete or partial) or stable disease lasting ≥6 months while on platinum-based therapy, or Platinum-free interval (PFI) ≥6 months from the end of the last platinum-containing regimen to documented progression/relapse.
6. Estimated life expectancy ≥3 months.
7. At least one measurable lesion per RECIST 1.1 on CT/MRI; evidence of metastatic disease (soft-tissue and/or bone lesions) is required.
8. Willing to provide archived tumour tissue (core biopsy or excision) or fresh biopsy/blood for biomarker analyses.
9. Adequate organ function within 14 days (7 days for liver enzymes) before first dose:

   Absolute neutrophil count ≥1.5 × 10⁹/L Platelets ≥100 × 10⁹/L Haemoglobin ≥80 g/L Total bilirubin ≤1.5 × upper limit of normal (ULN) ALT & AST ≤2.5 × ULN (≤5 × ULN if liver metastases present) Serum creatinine ≤1.25 × ULN and calculated creatinine clearance ≥60 mL/min
10. Toxicities from prior anti-cancer therapy resolved to Grade ≤1 per NCI-CTCAE v5.0 (except alopecia or other stable chronic toxicities deemed tolerable by the investigator).
11. Participants of reproductive potential and their partners must agree to use highly effective contraception from 30 days before the first dose until 120 days after the last dose of fluzoparib.
12. Signed written informed consent prior to any study-specific procedures.

Exclusion Criteria:

1. Known hypersensitivity to fluzoparib or any of its excipients.
2. Prior treatment with any PARP inhibitor.
3. Use of strong CYP3A4 inhibitors within 14 days or strong CYP3A4 inducers within 28 days before first dose.
4. Wash-out interval <4 weeks from any prior anti-cancer therapy (chemotherapy, radiotherapy, surgery, targeted therapy, immunotherapy) to first dose.
5. Planned anti-cancer therapy other than study drug during the trial period.
6. Severe bone complications from bone metastases (uncontrolled pain, impending pathological fracture, or spinal cord compression within 6 months or judged likely to occur).
7. Symptomatic or untreated brain metastases, leptomeningeal disease, spinal cord compression, or primary CNS tumors. (Stable brain metastases treated ≥28 days prior to first dose, without steroids and with confirmatory imaging showing no hemorrhage, may be allowed at investigator's discretion.)
8. Active autoimmune disease requiring systemic therapy within the past 2 years.
9. Recovery from major surgery under general anesthesia or severe trauma <14 days before start of study treatment.
10. Active hepatitis B (HBsAg positive and HBV DNA ≥500 IU/mL) or hepatitis C (anti-HCV positive and HCV RNA >ULN).
11. Untreated CNS metastases.
12. History of immunodeficiency (including HIV positive), congenital or acquired, or prior solid-organ transplant.
13. Other malignancies within 5 years except adequately treated carcinoma in situ or indolent tumors judged by the investigator to have low risk of recurrence.
14. Alcohol abuse (>14 units/week) or drug abuse; inability to stop smoking (>10 cigarettes/day), nicotine products, grapefruit juice, or excessive caffeine/tea during the study.
15. History of non-infectious pneumonitis requiring steroids or current pneumonitis.
16. Clinically significant ECG abnormalities, including QTcF >470 ms in females (QTc calculated with Fredericia's formula).
17. Conditions that could impair oral absorption: inability to swallow, active GI disease, bowel obstruction, inflammatory bowel disease, chronic diarrhea, short-bowel syndrome, or major upper-GI surgery (e.g., gastrectomy).
18. Active infection or unexplained fever >38.5 °C on screening or day 1 (tumor fever allowed if investigator judges stable).
19. Uncontrolled chronic systemic diseases (severe pulmonary, hepatic, renal, or cardiac).
20. Thyroid function abnormalities (TSH, FT3, FT4) deemed clinically significant by the investigator.
21. Bleeding diathesis: active peptic ulcer with positive fecal occult blood (FOB ++), melena or hematemesis within 2 months, or any condition predisposing to GI hemorrhage; gastric ulcer-type tumor without resection and judged at high risk of major bleeding; on thrombolytic/anticoagulant therapy that cannot be safely interrupted.
22. Urinalysis ≥++ proteinuria confirmed by 24-h urine protein >1.0 g.
23. Arterial or venous thrombo-embolic events (stroke, TIA, DVT, PE) within 6 months before screening.
24. Active tuberculosis or acute infection requiring anti-infective therapy.
25. Live-vaccine administration within 30 days before planned first dose.
26. Additional exclusion: Any severe concomitant condition that, in the investigator's opinion, could compromise patient safety or interfere with study compliance (e.g., uncontrolled diabetes, thyroid disorders, psychiatric illness).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From first dose of fluzoparib until disease progression or death, assessed every 6 weeks (2 cycles), up to approximately 12 months
  Time from first fluzoparib dose to first radiological disease progression (RECIST 1.1) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Second progression-free survival (PFS2) | From first fluzoparib dose until the above events, assessed every 6 weeks while on study and subsequently, up to approximately 24 months.
  Time from first dose of fluzoparib to the earliest of: radiological progression on next-line therapy, start of non-protocol anti-cancer treatment, or death from any cause.
Duration of response (DoR) | From first CR/PR documentation until progression or death, assessed every 6 weeks while on fluzoparib, up to approximately 24 months.
  Time from first documented complete or partial response (CR/PR) to subsequent radiological disease progression (RECIST 1.1) or death from any cause, whichever occurs first, among patients who achieved CR/PR
Disease control rate (DCR) | From first dose of fluzoparib until the 6-week tumor assessment, up to approximately 2 months.
  Proportion of participants achieving complete response, partial response, or stable disease (CR + PR + SD) lasting ≥ 6 weeks, assessed by RECIST 1.1
Overall survival (OS) | From first fluzoparib dose until death, assessed up to approximately 36 months.
  Time from first dose of fluzoparib to death from any cause.
Incidence and severity of adverse events (AE) | From first fluzoparib dose up to 30 days after last dose, assessed throughout the study and during follow-up, expected up to approximately 36 months.
  All adverse events will be recorded from first dose of fluzoparib until 30 days after last dose, graded by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No